CLINICAL TRIAL: NCT03402269
Title: Treatment of Pediatric Mid-shaft Clavicle Fractures: A Prospective, Observational Study
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00066019
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Clavicle Fracture; Adolescent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents with displaced clavicle fractures: Adolescents (11 to 17 years old) with displaced clavicle fractures will be enrolled in this study.
  Interventions: Other: Clavicle fracture injury- observation

INTERVENTIONS:
Other: Clavicle fracture injury- observation — The study is an observational study with assessments at 1 month, 3 months, 6 months and 1 year following injury. Assessments include range of motion, strength, patient reported outcomes and radiographic healing

SUMMARY:
Clavicle fractures in children are common. Typical treatment includes nonoperative treatment with a sling. Operative treatment is usually limited to open, unstable, fractures with either epidermal risks or neurovascular compromise. Orthopaedic literature has many studies that report the need for additional research for this prevalent fracture. This is an observational study evaluating the functional and patient reported outcomes of displaced clavicle fractures in adolescents. The results from this study will help the orthopedist understand the expected outcomes for a given pediatric patient with a clavicle fracture.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years old with fractures of the middle third of the clavicle
* Displaced 100% the width of the clavicle or shortened 1 centimeter
* Operative and non-operative treated clavicles will be eligible for enrollment

Exclusion Criteria:

* Open clavicle fractures
* Ipsilateral shoulder injuries
* Fractures involving the lateral ligaments or the sternoclavicular joint
* Bilateral clavicle fractures
* Pathologic fractures
* Refractures
* Fractures with neurovascular compromise
* Displaced fractures with impending skin compromise
* If there has been more than 21 days between injury and enrollment
* Patients with cognitive disabilities that inhibit the completion of the questionnaires

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 11-17 years old with displaced fractures of the middle third of the clavicle
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Range of motion | at 1 year post injury
  Range of motion measured by goniometer
Radiographic healing | at 1 year post injury
  Radiographic evidence of healing on 3 of 4 cortices

SECONDARY OUTCOMES:
QuickDash | at 3 months, 6 months and 12 months
  QuickDash Outcome Measure- measuring patient reported disability of arm, shoulder and hand
PODCI | at 3 months, 6 months and 12 months
  Adolescent Pediatric Outcomes Data Collection Instrument - measuring patient reported outcomes in a pediatric population

OTHER OUTCOMES:
Strength Measurements | 6 months and 12 months
  Upper extremity strength measurements, measured by dynamometer (forward flexion, abduction, and external rotation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Bray, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Hospital System, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD

DOCUMENTS (1):
  • Informed Consent Form (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03402269/ICF_000.pdf